CLINICAL TRIAL: NCT06322654
Title: A Head-to-head Study Comparing the Functional Value of Two Models of Robotically Assisted Rehabilitation in SMA Patients: Single-center, Randomized, Single-blinded, Comparative Study of a Robotically Active Verticalization Model Versus Robotically Assisted Locomotion Model
Brief Title: A Head-to-head Study Comparing the Functional Value of Two Models of Robotically Assisted Rehabilitation in SMA (Spinal Muscular Atrophy) Patients
Acronym: SMArt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wiktor Dega University Orthopedic and Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/ABM/01/00004/P/02
Record Dates: First submitted 2024-01-26; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: SMA
Keywords: SMA; Robotically-assisted therapy; Robotically Assisted Locomotion; Robotically Assisted Verticalization

STUDY DESIGN:
Intervention Model Description: There are two research groups with 100 patients in each group.
  1. Experimental: Robotically Assisted Locomotion
  2. Comparison: Robotically Assisted Verticalization
Who Masked: Investigator
Masking Description: Patients and their parents will not be blinded by the nature of the therapeutic procedure used after random allocation to the treatment group. Study personnel will be divided into Blinded Team and Unblinded Team to ensure objectivity of the assessment of safety and effectiveness of both strategies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotically Assisted Locomotion (Experimental)
  Interventions: Procedure: Robotically Assisted Locomotion
- Robotically Assisted Verticalization (Active Comparator)
  Interventions: Procedure: Robotically Assisted Verticalization

INTERVENTIONS:
Procedure: Robotically Assisted Locomotion — * Motor control training
  * Locomotion and motor control training with elements of balance and coordination
  * Verticalization training: standing frame device and vibration platform
  * Cognitive therapy
  Arms: Robotically Assisted Locomotion
Procedure: Robotically Assisted Verticalization — * Motor control training
  * Verticalization training with Standard Frame Devices
  * Locomotion and motor control training with elements of balance and coordination
  * Cognitive therapy
  Arms: Robotically Assisted Verticalization

SUMMARY:
A head-to-head study comparing the functional value of two models of robotically assisted rehabilitation in patients with SMA. A single-center, randomized, single-blinded, comparative study of Robotically Assisted Verticalization versus Robotically Assisted Locomotion.

The objective of research:

The main goal of the project is to determine the optimal robotically assisted rehabilitation model for people with SMA depending on age and baseline functional status. The study consists of a head-to-head comparison of two rehabilitation models.

1. Research period: 4 years
2. Patients age: 0-21 y.o.
3. Group size: 200 patients (100 patients in each group)
4. Assignment of patients to study groups in a randomised manner

ELIGIBILITY:
Inclusion Criteria:

* Signing of informed consent to participate in the experiment by the participant or the participant's parent/legal guardian
* Diagnosis of SMA (spinal muscular atrophy 1-4) confirmed by genetic testing, symptomatic or pre-symptomatic
* Age between 0 and 21 years of age (will be determined on the day of starting participation in the project based on the date of birth)
* Treatment under a drug program for spinal muscular atrophy, provided that the patient has a diagnosis of spinal muscular atrophy at the date of eligibility.

Exclusion Criteria:

* Cardio-respiratory disorders requiring invasive ventilation
* Advanced osteoporosis with multiple fractures prior to treatment
* Functional deterioration during the rehabilitation process in the range of scales appropriately selected for the SMA type: Prechtl, HINE, CHOP-INTEND, HFMS, RULM
* Lack of cooperation with the therapist
* Other functional indications preventing exercise

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of patients using Children's Hospital Of Philadelphia Infant Test Of Neuromuscular Disorders, Revised Upper Limb Module, Hammersmith Functional Motor Scale | Through study completion, max. for 2.5 year every 6 months
Clinical assessment of patients using Balance test minimum 1 min., Self-walk test of at least 2 meters, 6-minute gait test, Up&Go test, 10 meters gait test, hip range of motion and muscle strength evaluation. | Through study completion, max. for 2.5 year every 6 months
Functional assessment of patients using GMFM (Gross Motor Function Measure) scale | Through study completion, max. for 2.5 year every 6 months
X-ray or ultrasound scan imaging assessment of the spine, hip joints and bone mineral density | Once per 1 year
Assessment of the quality of life of patients and their caregivers using Pediatric Quality of Life Inventory ver. 4.0 | Through study completion, max. for 2.5 year every 6 months

SECONDARY OUTCOMES:
Hospitalization during or between rehabilitations that take place each 6 months | Through study completion, max. for 2.5 year
Occurence of discomfort during therapy requiring abrupt interruption or significant modification | Through study completion, max. for 2.5 year every 6 months
Number of fractures | Through study completion, max. for 2.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Marek Jóźwiak, Principal Investigator — Wiktor Dega University Orthopedic and Rehabilitation Hospital
Locations (1):
- Wiktor Dega University Orthopedic and Rehabilitation Hospital, Poznan, Poland